CLINICAL TRIAL: NCT05240001
Title: Thulium Fiber Laser (TFL) Versus Holmium MOSES Laser Enucleation of the Prostate for Treatment of Benign Prostatic Hyperplasia (BPH): A Randomized Prospective Clinical Study
Brief Title: Thulium Fiber Laser (TFL) vs Holmium MOSES for Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Principal Investigator, Hazem Elmansy, Urologist, Thunder Bay Regional Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-775
Record Dates: First submitted 2022-01-07; First posted 2022-02-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium Fibre Laser (TFL) (Experimental): Patients randomized to this arm will undergo treatment using the TFL.
  Interventions: Device: Thulium Fibre Laser
- MOSES Holmium Laser (Experimental): Patients randomized to this arm will undergo treatment using the MOSES Holmium laser.
  Interventions: Device: MOSES Holmium Laser

INTERVENTIONS:
Device: Thulium Fibre Laser — Participants will undergo treatment using the TFL
  Arms: Thulium Fibre Laser (TFL)
Device: MOSES Holmium Laser — Participants will undergo treatment using the MOSES Holmium laser.
  Arms: MOSES Holmium Laser

SUMMARY:
Benign prostatic hyperplasia (BPH), the non-cancerous enlargement of the prostate, places pressure on the urethra and causes urination and bladder problems. Transurethral Resection of the Prostate (TURP) remains the gold standard treatment in most centres for BPH. However, morbidity after TURP is high, especially bleeding requiring blood transfusion and late postoperative bleeding.

Holmium laser enucleation of the prostate (HoLEP) is a safe and effective procedure which has demonstrated comparable results to TURP. HOLEP also offers patients the alternative of being treated endoscopically with minimal blood loss, short catheterization time, and decreased hospital stay. The main reason HoLEP has yet to become the new standard for treatment of symptomatic BPH is due the complexity of this procedure as compared to TURP. Furthermore, the HoLEP can be used with the MOSESTM system, a system that allows for more efficiency and ease of use of the HoLEP.

Thulium fiber laser (TFL) enucleation of the prostate is an emerging technology for endoscopic prostate enucleation that is notable for its high wavelength and pulsed mode of action. Recent studies have shown TFL enucleation of the prostate to be a safe and highly efficacious treatment modality for the management of large volume (> 80 cm3) glands in BPH. Due to its novelty, further studies are needed to broaden the investigators' understanding of the TFL and comprehend the full implications and benefits of this new technology, as well its limitations.

The aim of this study is to whether Thulium Fiber laser enucleation of the prostate (ThuFLEP) and Holmium laser enucleation using MOSES™ (M-HoLEP) have comparable length of hospital stay, as well as intraoperative and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males over 50 years of age at the time of enrollment
2. Referred to urology for refractory LUTS or urinary retention secondary to BPH
3. Failed medical (non-surgical) treatment
4. Prostate size on preoperative TRUS of≥80 ml
5. IPSS >15 and QOL score ≥3 and Qmax <15 ml/sec
6. Written informed consent to participate in the study
7. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Previous surgical treatment for BPH
2. History of prostate cancer
3. Prostate size < 80 mL
4. History of urethral stenosis or its management
5. Known or suspected neurogenic bladder
6. Participants with active urinary tract infection until appropriately treated
7. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study
8. Participants who lack the capacity, or cannot speak English, in order to provide free and informed written consent

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Length of stay in the hospital | within 6 hours

SECONDARY OUTCOMES:
Incidence of bleeding | Intra-Op
Incidence of blood transfusion | Intra-Op
Operative time | Intra-Op
  Including laser use time
International Prostate Symptom Score | 1,3,6,12 months post-op
  Eight questions (seven concerning urinary symptoms and one concerning quality of life), responses range from 0 (better outcome) to 5 (worse outcome), with total score ranging from 0 to 35.
Quality of Life (QOL) as scored on the International Prostate Symptom Score (IPSS) | 1,3,6,12 months post-op
  Response to the last question on the IPSS:
  "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" Response ranging from 'Delighted' to 'Terrible'.
Peak flow rate | 1,3,6,12 months post-op
  Qmax
Post-void residual | 1,3,6,12 months post-op
  PVR
Prostate specific antigen | 1,3,6,12 months post-op
  PSA
Change in size | 6 months
  Assessed by TRUS
Time to Catheter Removal | within 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, MD, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No